CLINICAL TRIAL: NCT02384811
Title: Phase II Study of Extensive Clinical Target Volumes in Postoperative Radiotherapy for Esophageal
Brief Title: Phase II Study of Extensive Clinical Target Volumes in Postoperative Radiotherapy for Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jiaqing Xiang, director, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-86-882
Record Dates: First submitted 2015-03-02; First posted 2015-03-10 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal squamous cell carcinoma; postoperative radiotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation group (Experimental): Radiation therapy
  Interventions: Radiation: radiation

INTERVENTIONS:
Radiation: radiation — A total dose of 40Gy will be delivered in 20 fractions at 2.0Gy/fraction, 5 fractions per week in 4 weeks.
  The CTV encompassed the bilateral supraclavicular region, all mediastinal lymph nodes, the anastomosis site, and the left gastric and Celiac nodes.

SUMMARY:
The primary object of this trial is to evaluate the 2-year local control rate adding extensive clinical target volumes in postoperative radiotherapy for esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Joined the study voluntarily and signed informed consent form;
* Age 18-75；ECOG 0-2
* Esophageal squamous cell carcinoma , radical surgery ≤3 months,R0 resection. The operative incision healed well.
* T3-4N0M0, T1-4N1-3M0 (according to AJCC2009)
* No radiotherapy, chemotherapy or other treatments pre(post)surgery
* PS ECOG 0-2
* Life expectancy of more than 3 months
* Hemoglobin(Hb)≥9 g/dL • WBC≥3x109/L, Neutrophils (ANC )≥1.5x109/L • platelet count (Pt) ≥100x 109/L • Hepatic function: ALAT and ASAT < 2.5 x ULN, TBIL<1.5 x ULN • Renal function: creatinine < 1.5 x ULN
* No immuno-deficiency
* Use of an effective contraceptive for adults to prevent pregnancy.

Exclusion Criteria:

* Complete esophageal obstruction after surgery, Esophageal perforation, Haematemesis
* Other malignant tumors, except for skin basal cell carcinoma, or cervical carcinoma in situ, who survived with no evidence disease for over 3 years
* Participation in other interventional clinical trials within 30 days
* Pregnant or breast-feeding women or people during the birth-period who refused to take contraceptives
* Drug addiction, Alcoholism or AIDS
* Uncontrolled seizures or psychiatric diseases, loss of control over their own behavior
* Unsuitable to be enrolled in the trial in the opinion of the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Local control rate | 2 years

SECONDARY OUTCOMES:
Overall survival | 5 year
Safety: Frequencies of treatment-related adverse event categories by NCI-CTC | 3 months
  Frequencies of treatment-related adverse event categories by NCI-CTC including Esophagitis,Pneumonitis/Bronchitis,Skin reaction in radiation fields,Nausea/vomiting,Leucopenia,Thrombocytopenia,Anemia,Fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-qing Xiang, M.M, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Cancer hospital Fudan University, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Zhang X, Ai D, Wang J, Chen Y, Liu Q, Deng J, Yang H, Nie Y, Chen W, Zhao W, Zhao K. The Prognosis and Feasibility of Extensive Clinical Target Volume in Postoperative Radiotherapy for Esophageal Squamous Cell Carcinoma: A Phase II Clinical Trial. Front Oncol. 2021 Jul 2;11:669575. doi: 10.3389/fonc.2021.669575. eCollection 2021. PMID 34295813